CLINICAL TRIAL: NCT04381910
Title: A Phase Ⅱ Study Evaluate the Efficacy and Safety of LY01610（Irinotecan Hydrochloride Liposome Injection） in Patients With Small Cell Lung Cancer
Brief Title: Irinotecan Hydrochloride Liposome Injection (LY01610) For Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY01610/CT-CHN-202
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Small Cell Lung Cancer
Keywords: LY01610; Efficacy; Safety; Irinotecan Hydrochloride Liposome Injection; Second-Line Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LY01610 (Experimental): LY01610(Irinotecan Hydrochloride Liposome Injection),Patients were enrolled in one to three cohorts to receive LY01610 every 2 weeks, initial 30 subjects will be included in each cohort and the number of the cases could be adjusted. Subjects will receive LY01610 start with 60 mg/m2 every 2 weeks，when the sixth subjects of the current cohort completed 14 days safety observation of the first LY01610 administration, the investigators will evaluate the ongoing dose tolerance. If the investigator and the sponsor jointly believe that other doses can provide greater potential benefits for patients while ensuring safety and benefit, other appropriate cohorts could be explored (such as 80, 90 and 100 mg/m2, etc.) Subjects will receive the LY01610 monotherapy until occurrence of progressive disease (PD), death, intolerable toxicity reaction, withdrawal of informed consent, conduct of other antitumor therapy or completion of the whole study.
  Interventions: Drug: LY01610( Irinotecan hydrochloride liposome injection )

INTERVENTIONS:
Drug: LY01610( Irinotecan hydrochloride liposome injection ) — LY01610 will be administered via intravenous infusion every 2 weeks on Day 1

SUMMARY:
This is a Multicenter, Non-randomized, Open Label, Multiple Dose, Multiple administration, Phase IIa Clinical Study Evaluating the Efficacy and Safety of LY01610 in Patients with Extensive-stage Small Cell Lung Cancer that Progressed after first-line Antitumor Therapy.

DETAILED DESCRIPTION:
The objectives are to evaluate the efficacy and safety of LY01610 in subjects with extensive small cell lung cancer that progressed after first-line antitumor therapy.

Patients were enrolled in one to three cohorts to receive LY01610 every 2 weeks, initial 30 subjects will be included in each cohort and the number of the cases could be adjusted. Subjects will receive LY01610 start with 60 mg/m2 every 2 weeks，when the sixth subjects of the current cohort completed 14 days safety observation of the first LY01610 administration, the investigators will evaluate the ongoing dose tolerance. If the investigator and the sponsor jointly believe that other doses can provide greater potential benefits for patients while ensuring safety and benefit, other appropriate cohorts could be explored (such as 80, 90 and 100 mg/m2, etc.) Subjects will receive the LY01610 monotherapy until occurrence of progressive disease (PD), death, intolerable toxicity reaction, withdrawal of informed consent, conduct of other antitumor therapy or completion of the whole study.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female patients aged 18 to 70 years (18 years and 70 years are inclusive).

  2.Histologically or cytologically confirmed extensive small cell lung cancer. 3.Disease progression or recurrence after one prior systematic anti-tumor treatment regimen (including platinum-containing chemotherapy, etc.; with or without radiotherapy).

  4.The patient should have at least one measurable lesion (according to RECIST 1.1 criteria).

  5.Life expectancy ≥3 months. 6.The Eastern Cooperative Oncology Group (ECOG) performance status score is between 0 to 1 point.

  7.Laboratory results during screening:
  * Hematology：Absolute neutrophil count ≥ 1.5× 109/L, platelet count≥ 100× 109/L and hemoglobin≥ 90 g/L.
  * Liver function: Total bilirubin <1.5×upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN for the subjects without liver metastasis; ALT and AST≤5×ULN for the subjects with liver metastasis.
  * Kidney function: Serum creatinine ≤ 1.5 ×ULN or creatinine clearance rate ≥ 50 mL/min.
  * Coagulative function: Prothrombin time - international standardized ratio（PT-INR） <1.5.

    8.The subject has voluntarily signed the written informed consent form (ICF) and can comply with the study protocol.

    9.The female subjects and male subjects of childbearing age and the partners of the male subjects agree to take reliable contraceptive measures (such as abstinence, sterilizing operation, contraceptives, injection of the contraceptive drug medroxyprogesterone acetate or subdermal implant of contraceptives) during the study period and within 6 months after infusion of the study drugs.

Exclusion Criteria:

* 1.Patients with the symptomatic brain metastasis, meningeal metastases, spinal cord tumor invasion, spinal cord compression. Patients with superior vena cava syndrome, obstructive atelectasis and bone metastasis who have local symptoms, which may require radiotherapy / surgery / endoscopic treatment / interventional treatment and other non-medical treatment.

  2.Patients have other malignant tumors within 5 years(except for cured stage ⅠB or lower cervical cancer, non-invasive basal cell or squamous cell skin cancer) 3.Uncontrolled massive hydrothorax, ascites and pericardial effusion. 4.Patients have history of deep vein thrombosis or pulmonary embolism. 5.The patient with persistent or active infection signs which need intravenous injection of antibiotics.

  6.Medical history of the following diseases within 6 months: myocardial infarction, unstable angina pectoris, coronary revascularization, cardiac dysfunction (New York heart association (NYHA) grade ≥ II), severe unstable ventricular arrhythmia or arrhythmias that need to be treated at the time of screening.

  7.The patient with Active hepatitis B: hepatitis B surface antigen (HBsAg) positive and the peripheral blood hepatitis B virus DNA (HBV DNA)titer ≥1× 103 copies/mL or 200 IU/ml. The subject is eligible to be enrolled if HBsAg is positive and peripheral blood HBV DNA titer <1×103 copies/mL or 200 IU/ml and the investigator considers that the subject is at the stable stage of chronic hepatitis and the risk will not be increased for the subject. The patient with hepatitis C virus (HCV) antibody positive, human immunodeficiency virus (HIV) antibody positive and active syphilis infection.

  8.Patients have severe gastrointestinal disorders (such as gastrointestinal bleeding, infection, chronic enteritis, obstruction, or diarrhea with CTCAE grade 1 or higher) at the time of screening.

  9.Patients with medical history of neuropathy or mental disorder (including epilepsy or dementia).

  10.Patients have been or are suffering from bronchial asthma, interstitial lung disease or active hemoptysis within 6 months.

  11.Patients with primary diseases of other major organs (such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system or metabolic endocrine system) and the investigators believe that it is not suitable for enrollment, or for other reasons the investigators don't think that suitable for inclusion.

  12.Patients who have previous treatment with irinotecan or immunotherapy. 13.Known hypersensitivity to any of the components of irinotecan liposome injection, other structurally similar compounds (such as camptothecins), or other liposomal products.

  14.Patients have participated in other pharmaceutical clinical trial within one month before screening.

  15.Patients have received systemic antitumor therapy such as radiation, chemotherapy, immunotherapy or other treatments within 4 weeks prior to start of therapy.

  16.Patients have received live or attenuated vaccines within one month prior to the screening.

  17.Use of strong CYP3A4 inducers (phenytoin or carbamazepine, barbiturates, rifampin, rifabutin or rifapentine, hypericum perforatum, etc) during or within 14 days prior to starting study medication.

  18.Use of strong CYP3A4 inhibitors (clarithromycin, ketoconazole or itraconazole, indinavir, lopinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telaprevir,voriconazole, etc) during or within 14 days prior to starting study medication. 19.Use of strong UGT1A1 inhibitors during or within 14 days prior to starting study medication (atazanavir, gemfibrozil, indinavir, etc.).

  20.Patients who are taking or may take drugs that reduce cholinesterase activity or choline drugs (neostigmine, lissamine, acetylcholine, etc.).

  21.Patients may used the skeletal muscle relaxation drugs (such as succinylcholine) during the trial.

  22.The patient who has drug and/or alcohol abuse. 23.Pregnant or lactating women. 24.Patients who did not take contraceptive measures during the trial. 25.Other circumstances which are considered by the investigator that the subject is unsuitable to be enrolled.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
Duration of Response(DoR) | from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
Progression Free Survival(PFS) | from the date of randomisation to the date of disease progression or death up to 12 months from randomisation of the last subject
Overall Survival(OS) | from the date of randomisation to the date of death up to 12 months from randomisation of the last subject

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, Professor, Principal Investigator — Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No